CLINICAL TRIAL: NCT06117163
Title: Integration of a Collaborative Care Model for Mental Health Services Into HIV Care for Pregnant and Postpartum Women in Kenya (the Tunawiri Study)
Brief Title: Integrated Mental Health Care for Pregnant Women With HIV in Kenya: The Tunawiri Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: University of North Carolina, Chapel Hill (Other); Kenya Medical Research Institute (Other); University of Alabama at Birmingham (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 23-0498
Record Dates: First submitted 2023-10-30; First posted 2023-11-03 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Human Immunodeficiency Virus; Mental Disorder
Keywords: HIV transmission; Prevention of Mother to Child Transmission; Linkage to care; Retention in care; Antiretroviral therapy adherence; Infant Health; Maternal CD4/viral loads; Early infant diagnosis; Acceptability of interventions; Vertical transmission; Mental Health; The Collaborative Care Model; Problem Solving Therapy; Stigma
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Mental Disorders; Psychological Well-Being; Social Stigma

STUDY DESIGN:
Intervention Model Description: A type 2 hybrid effectiveness-implementation trial with a stepped-wedge design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Collaborative Care Model (CCM) (Experimental): The investigators propose a CCM called Tunawiri, meaning "thrive" in Kiswahili, that will be integrated within an existing multidisciplinary team of clinicians, mentor mothers, and other clinic staff in Kenyan antenatal care clinics. CCM includes: 1) clinic-level sensitization and integration, 2) Screening for CMD including anxiety, depression and trauma symptoms, 3) Problem-solving type cognitive behavioral therapy delivered by lay health workers, 4) Decision Support and monitoring via an Electronic Health Registry, and 5) Psychiatrist case review and nurse-managed mental health medication.
  Interventions: Behavioral: Collaborative Care Model

INTERVENTIONS:
Behavioral: Collaborative Care Model — The investigators propose a CCM called Tunawiri, meaning "thrive" in Kiswahili, that will be integrated within an existing multidisciplinary team of clinicians, mentor mothers, and other clinic staff in Kenyan antenatal care clinics. CCM includes: 1) clinic-level sensitization and integration, 2) Screening for CMD including anxiety, depression, and trauma symptoms, 3) Problem-solving type cognitive behavioral therapy delivered by lay health workers, 4) Decision Support and monitoring via an Electronic Health Registry, and 5) Psychiatrist case review and nurse-managed mental health medication.
  Other Names: Tunawiri model

SUMMARY:
This study seeks to improve mental health, pregnancy, and HIV outcomes among pregnant and postpartum women living with HIV with common mental health disorders in Kenya. The investigators will tailor a collaborative care model for peripartum women with HIV experiencing mental health symptoms and evaluate its impact on participants' mental health, antenatal, and HIV care outcomes. The investigators will actively engage key stakeholders throughout the process and assess scalability and sustainability through multi-method approaches. This study will contribute to the overall goal of achieving optimal health outcomes for women living with HIV and their families in sub-Saharan Africa.

DETAILED DESCRIPTION:
Common mental disorders (CMD) of depression and anxiety are prevalent and largely untreated among Kenyan pregnant and postpartum women living with HIV (PPWH). CMD lead to poor maternal and child health outcomes and contribute to lack of HIV care engagement and virologic failure in PPWH. While efficacious treatments for CMD exist, scaling treatment within routine health care in low- and middle-income (LMIC) settings will require stakeholder engagement and both effectiveness and implementation data to inform scale up and sustainability. The study team has integrated other efficacious interventions into antenatal (ANC) and HIV care in Kenya. The investigators now propose to integrate proven mental health services using a collaborative care model, combined with a low intensity evidence-based intervention (problem solving therapy), while targeting known social determinants of HIV-related health for PPWH (stigma and IPV). Building on the current multidisciplinary approach for HIV care in Kenya, the proposed Collaborative Care Model (CCM) will utilize existing peer mentor mothers, non-specialist behavioral care managers, and psychiatric nurses; and will incorporate a consultant psychiatrist into the ANC/HIV care team. Guided by the EPIS (Exploration-Preparation-Implementation-Sustainment) framework, the overall study goal is to integrate collaborative care for perinatal CMD within routine ANC/HIV services in Kenya, assess the costs and cost-effectiveness of this approach, and work with policy and decision makers to determine key considerations for scale-up. Specifically, in Aim 1, the investigators will identify contextual barriers and facilitators to refine an optimal integration model for delivering collaborative care model using multimethod data collection (focus groups with providers, in-depth interviews with key informants, and a clinic readiness checklist). A workshop with the study Advisory Board comprising of both county and national level stakeholders, will allow investigators to translate findings into a locally relevant CCM. In Aim 2, the investigators will test CCM in antenatal care for PPWH in a hybrid type 2 implementation-effectiveness trial using a stepped wedge design at 15 primary health care facilities in southwestern Kenya. The investigators will introduce CCM care for PPWH diagnosed with CMD during antenatal care. The co-primary health outcomes at 12 months postpartum will be (1) recovery from depression or anxiety symptoms in PPWH, and (2) proportion PPWH with sustained viral suppression and retention in HIV care. Key implementation outcomes are feasibility and acceptability. Finally, in Aim 3, the investigators will refine CCM implementation strategies through cost-effectiveness and dissemination research. The investigators will carry out costing and cost-effectiveness analysis and invite policy and decision-makers to participate in a nominal group technique process to elucidate factors for further scale up and sustainment of the CCM approach. Findings from this study will guide the development of a scalable model adaptable to other LMIC settings, contributing to global HIV and maternal health goals while addressing the burden of untreated CMD.

ELIGIBILITY:
Inclusion Criteria:

* pregnant woman living with HIV attending an antenatal clinic in southwestern Kenya
* screening positive for probable common mental disorders
* living in catchment area of study facility.
* on/initiating ART
* >15 years of age

Exclusion Criteria:

* imminent plans of suicide
* severe impairment due to severe mental, neurological or substance use disorders.

Min Age: 15 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 900 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2028-05-31 (Estimated)

PRIMARY OUTCOMES:
Recovery of women from depression | Baseline, 6 months postpartum, 12 months postpartum
  Depression score is calculated and severity assessed through a survey utilizing the Patient Health Questionnaire Depression Scale (PHQ-9). PHQ-9 score is obtained by adding a score for each question (total points). A total score of 0-4 suggests none to minimal depression severity, a score of 5-9 mild depression severity, a score of 10-19 moderate depression severity, and a score of 20-27 severe depression. Recovery from depression of pregnant and postpartum women living with HIV will be assessed as the change of a total PHQ-9 score from >10 points to equal or less 10 points between baseline and 12 months postpartum.
Recovery of women from anxiety | Baseline, 6 months postpartum, 12 months postpartum
  Anxiety score is calculated and severity assessed through a survey utilizing the Generalized Anxiety Disorder 7-item (GAD-7). GAD-7 score is obtained by adding a score for each question (total points). A total score of 0-4 suggests none to minimal anxiety severity, a score of 5-9 mild anxiety severity, a score of 10-14 moderate anxiety severity, and a score of 15-21 severe anxiety. Recovery from the anxiety of pregnant and postpartum women living with HIV will be assessed as the change of a total GAD-7 score from >10 points to equal or less 10 points between baseline and 12 months postpartum.
Change in the proportion of women with combined retention and treatment success outcome | Baseline, 6 months postpartum, 12 months postpartum
  The change in the proportion of women with the combined outcome of HIV care retention (didn't miss any HIV care appointment by 14 or more days) and a suppressed HIV RNA (<400 copies/ml) among pregnant and postpartum women living with HIV assessed through medical records between baseline, 6 months postpartum, and 12 months postpartum.

SECONDARY OUTCOMES:
Infant weight at birth | Birth
  A birth weight, measured in grams, and based on medical records, and categorized into normal weight (equal or more than 2500 grams at birth), low birth weight (<2500 grams at birth), very low birth weight (<1,500 grams at birth), and extremely low birth weight (<1,000 grams at birth).
Proportion of women with preterm delivery of women who experienced adverse pregnancy outcomes | Birth
  The proportion of women who experienced a preterm delivery, measured as delivery <37 weeks of pregnancy) based on medical records.
Result of infant HIV test | Birth, 6 weeks, 6 months, 12 months
  Result of infant HIV test at birth, 6 weeks, 6 months, and 12 months, assessed through medical records and categorized into HIV positive or HIV negative.
Infant retention in care | Birth, 6 weeks, 6 months, 12 months
  Continuous visit adherence from birth through 12 months after birth (no missed clinic/pharmacy visit >14 days) assessed through medical records.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Abuogi, MD, MSc, Principal Investigator — University of Colorado, Denver
Locations (1):
- Kenya Medical Research Institute, Nairobi, Kenya